CLINICAL TRIAL: NCT00213382
Title: Cortical Pharyngeal Area: Excitability, Facilitation and Plasticity in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Other Study IDs: 2003/031/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: swallowing; ventilation; pressure; EMG; cortical magnetic stimulation; Brain Mapping
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aims of this study are in four experimental sessions. The aims are:

* to characterize the excitability of the cortical pharyngeal area with pharyngeal pressure and electromyograms (EMGs), at rest, in awake healthy subjects;
* to study its facilitation by inspiration and deglutition; and
* to study its plasticity by respiration and swallowing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Eric Verin, MD, PhD, Principal Investigator — University Hospital, Rouen; Eric Verin, MD, PhD, Principal Investigator — University CHU Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France